CLINICAL TRIAL: NCT06078254
Title: Accuracy, Senstivity and Specificity of Lung Ultrasound in Comparison to CT Chest for Early Detection of ARDS and Pneumonia in Patients With Chest Trauma
Brief Title: Senstivity and Specificity of Lung Ultrasound for Early Detection of ARDS in Patients With Chest Trauma
Status: Recruiting | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: Ultrasound in chest trauma
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Chest Trauma
MeSH Terms: conditions — Thoracic Injuries | interventions — Ultrasonography; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: ULTRASOUND — Ultrasound and CT chest for all patients
  Other Names: COMPUTERIZED TOMOGRAPHY

SUMMARY:
The aim of this study is to evaluate the accuracy, sensitivity and specificity of lung ultrasound in early detection of ARDS and Pneumonia in comparison to CT chest in patients with chest trauma. Also, we aim at finding any pulmonary complications and its correlation to development of ARDS and pneumonia in patients with chest trauma.

DETAILED DESCRIPTION:
Thoracic trauma has significant morbidity and mortality. It is the fourth most common trauma site after the head, abdomen, pelvis and extremities.

Thoracic trauma is one of the critical injury mechanisms in multiply injured trauma victims. Although these patients present a plethora of potential structural damages to vital organs, it remains debated which injuries actually influence outcome and thereby should be addressed initially.

Routine tests for chest injuries include chest X-rays and computed tomography (CT) scans. Chest X-rays are available but are insufficiently sensitive for chest trauma. Multi-detector CT is now considered the gold standard imaging tool in the emergency department; however, it is not applicable for unstable patients and is unavailable in intensive care units, so patient transport to radiology departments is required. This technique also exposes patients to high doses of ionizing radiation.

In thoracic trauma cases, ultrasonography of the lungs is valuable for evaluating various chest diseases, including chest wall hematoma and fractures, pleural cavity involvement with pleural effusion, hemothorax, and pneumothorax, and pericardial cavity involvement with hemopericardium.

The ultrasound can also assess the reduce in lung aeration in acute diseases by changing the lung surface and generating distinct patterns as in pulmonary contusions and compression atelectasis.

In pneumothorax cases, the major criterion for ultrasound diagnosis is the absence of lung sliding during a dynamic examination, as well as the absence of a pleural gap and lung point, which is the transitional area between the breath-dependent, moving lung and the pleural air column in cases of partial pneumothorax with incomplete lung collapse.

Lung contusion is the most frequent thoracic injury in blunt chest trauma and it is associated with increased morbidity and mortality. Direct damage of the lung tissue causes both local and systemic inflammatory responses that can lead to acute respiratory distress syndrome (ARDS) and multiple organ failure. The initial size of the lung contusion seems to play a key role in these mechanisms.Several CT scan studies have shown that initial lung contusion volume is predictive of the development of subsequent ARDS.

Ultrasounds aids in pleural effusion detection, even if minimal. Ultrasound can assess and quantify the amount of effusion, and characterize its internal complexity, such as septations, exudative effusion, fibrin strands, and echogenic pleural effusion.

ELIGIBILITY:
Inclusion Criteria:

* All ICU patients who got admitted to critical care department with chest trauma.

Exclusion Criteria:

* Pediatric patients aged less than 18 years old.
* Any patients have previous lung disease like (IPF, lung cancer, respiratory failure and pulmonary hypertension).
* Pregnant females at any gestational age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who admitted to critical area with chest trauma will perform both CT chest and lung ultrasound and will be followed up by ultrasound to detect any pulmonary complication and early detection of ARDS and pneumonia.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of accuracy ,sensitivity and specificity of lung ultrasound in early detection of acute respiratory distress syndrome and pneumonia in patients with chest trauma. | 18 MONTHS
  Evaluation of accuracy ,sensitivity and specificity of lung ultrasound in early detection of acute respiratory distress syndrome and pneumonia in patients with chest trauma.

SECONDARY OUTCOMES:
Correlation between occurrence of different pulmonary complications due to chest trauma and development of ARDS and pneumonia in patients with chest trauma. | 18 MONTHS
  Correlation between occurrence of different pulmonary complications due to chest trauma and development of ARDS and pneumonia in patients with chest trauma.

CONTACTS AND LOCATIONS:
Overall Officials: Omar M. Taha Elsafty, professor, Study Chair — Ain Shams University; Kareem Y. Kamal Hakim, professor, Study Director — Ain Shams University; Amr G. Sharaf, MD, Study Director — Ain Shams University; Eman M. Hesham Elshaer, MD, Study Director — Ain Shams University
Locations (1):
- AinShams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dogrul BN, Kiliccalan I, Asci ES, Peker SC. Blunt trauma related chest wall and pulmonary injuries: An overview. Chin J Traumatol. 2020 Jun;23(3):125-138. doi: 10.1016/j.cjtee.2020.04.003. Epub 2020 Apr 20. PMID 32417043
- [Background] Ferrer M, Difrancesco LF, Liapikou A, Rinaudo M, Carbonara M, Li Bassi G, Gabarrus A, Torres A. Polymicrobial intensive care unit-acquired pneumonia: prevalence, microbiology and outcome. Crit Care. 2015 Dec 23;19:450. doi: 10.1186/s13054-015-1165-5. PMID 26703094
- [Background] Francone M, Iafrate F, Masci GM, Coco S, Cilia F, Manganaro L, Panebianco V, Andreoli C, Colaiacomo MC, Zingaropoli MA, Ciardi MR, Mastroianni CM, Pugliese F, Alessandri F, Turriziani O, Ricci P, Catalano C. Chest CT score in COVID-19 patients: correlation with disease severity and short-term prognosis. Eur Radiol. 2020 Dec;30(12):6808-6817. doi: 10.1007/s00330-020-07033-y. Epub 2020 Jul 4. PMID 32623505
- [Background] Mardani P, Moayedi Rad M, Paydar S, Amirian A, Shahriarirad R, Erfani A, Ranjbar K. Evaluation of Lung Contusion, Associated Injuries, and Outcome in a Major Trauma Center in Shiraz, Southern Iran. Emerg Med Int. 2021 Apr 22;2021:3789132. doi: 10.1155/2021/3789132. eCollection 2021. PMID 33976939
- [Background] Pan F, Ye T, Sun P, Gui S, Liang B, Li L, Zheng D, Wang J, Hesketh RL, Yang L, Zheng C. Time Course of Lung Changes at Chest CT during Recovery from Coronavirus Disease 2019 (COVID-19). Radiology. 2020 Jun;295(3):715-721. doi: 10.1148/radiol.2020200370. Epub 2020 Feb 13. PMID 32053470
- [Background] Soni NJ, Franco R, Velez MI, Schnobrich D, Dancel R, Restrepo MI, Mayo PH. Ultrasound in the diagnosis and management of pleural effusions. J Hosp Med. 2015 Dec;10(12):811-6. doi: 10.1002/jhm.2434. Epub 2015 Jul 28. PMID 26218493
- [Background] Raghavendran K, Notter RH, Davidson BA, Helinski JD, Kunkel SL, Knight PR. Lung contusion: inflammatory mechanisms and interaction with other injuries. Shock. 2009 Aug;32(2):122-30. doi: 10.1097/SHK.0b013e31819c385c. PMID 19174738
- [Background] Hyllienmark P, Brattstrom O, Larsson E, Martling CR, Petersson J, Oldner A. High incidence of post-injury pneumonia in intensive care-treated trauma patients. Acta Anaesthesiol Scand. 2013 Aug;57(7):848-54. doi: 10.1111/aas.12111. Epub 2013 Mar 31. PMID 23550742